CLINICAL TRIAL: NCT05783999
Title: Role of Muscle Vibration in Improving the Sense of Fatigue in Patients With Multiple Sclerosis
Brief Title: Muscle Vibration and Fatigue in Patients With MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Roberta Cellini, MD, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VIBRATIPLA
Record Dates: First submitted 2023-03-14; First posted 2023-03-24 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard care + vibra plus (Experimental): patients will undergo treatment with the vibra plus device on top of traditional rehabilitation
  Interventions: Device: vibra plus
- Standard care (No Intervention): patients undergo a traditional rehabilitation program

INTERVENTIONS:
Device: vibra plus — the device is applied to the patient's lower limbs and generates an active flow of vibrations that may reduce fatigue
  Arms: standard care + vibra plus

SUMMARY:
Multiple Sclerosis is the most common cause of neurologic chronic disability in young adults. Fatigue is one of the principal symptom in this disease.

In the past it was demonstrated how, with appropriate frequencies and amplitude of vibration, it is possible both to select the activated afferents, and to determine the frequency of action potentials sent to the Central Nervous System.

The purpose of this study is to verify how the use of vibrations can induce positive effects on the mobility and postural control of patients with MS, as well as reduce fatigue.

The study is an interventional type. The subjects are undergoing to baseline examinations (T0) including 3D gait analysis (using a BTS system), stabilometric analysis, and a battery of neuropsychological assessments. Subsequently, eligible subjects are undergoing to intensive multidisciplinary training for a total of 5 sessions per week for 4 weeks, with a total of 20 treatment sessions. The experimental group receive additional vibration treatment. At the end of the treatment cycle (T1), the patients will undergo the same evaluation tests as at baseline. The Clinical and instrumental exams used for this study (as per normal clinical practice) are: Expanded Disability Status Scale (EDSS), Fatigue Severity Scale (FSS), Modified Fatigue Impact Scale (MFIS), Fatigue Scale for Motor and Cognitive Functions (FSMC), Borg Scale, Medical Research Council Scale (MRC), 6 minutes walking test.

The Psychological Assessment Battery used are: Multiple Sclerosis Quality of Life-54 (MSQOL-54) scale, Beck Depression Inventory-II, Coping Orientation to Problems Experienced (COPE).

Sample size: The sample consist of patients with MS admitted to the C.A.R.E.N. or Casazza facilities of the IRCCS Centro Neurolesi Bonino-Pulejo in Messina. Twenty eligible subjects recruited and treated with traditional rehabilitation approach plus vibrational therapy. The results will be compared to those obtained from a group of 20 patients who have undergone a traditional rehabilitation treatment without the application of vibrations and who will represent the control group.

DETAILED DESCRIPTION:
Multiple Sclerosis is the most common cause of neurologic chronic disability in young adults.

Fatigue is one of the principal symptom in this disease. Fatigue in a subject with MS is present every day, gets worse as the day progresses, with the heat and humidity, it is sudden and more severe than normal, it interferes with physical performance. Fatigue is prevalent in the MS population and is a significant health problem, negatively impacting activities of daily living, ability to work, social life and quality of life.

In 1963 it was demonstrated how mechanical vibration, applied to a single muscle, at suitable amplitudes and frequencies, was capable of selectively and differentially activating primary (Ia), secondary (IIb) or GTO spindle afferents, depending on the characteristics of the stimulus. So with appropriate frequencies and amplitude of vibration, it is possible both to select the activated afferents, and to determine the frequency of action potentials sent to the Central Nervous System. The purpose of this study is to verify how the use of vibrations can induce positive effects on the mobility and postural control of patients with MS, as well as reduce fatigue. The study is an interventional type. The subjects are undergoing to baseline examinations (T0) including 3D gait analysis (using a BTS system), stabilometric analysis, and a battery of neuropsychological assessments. Subsequently, eligible subjects are undergoing to intensive multidisciplinary training for a total of 5 sessions per week for 4 weeks, with a total of 20 treatment sessions. The experimental group receive additional vibration treatment. At the end of the treatment cycle (T1), the patients will undergo the same evaluation tests as at baseline. The Clinical and instrumental exams used for this study (as per normal clinical practice) are: Expanded Disability Status Scale (EDSS), Fatigue Severity Scale (FSS), Modified Fatigue Impact Scale (MFIS), Fatigue Scale for Motor and Cognitive Functions (FSMC), Borg Scale, Medical Research Council Scale (MRC), 6 minutes walking test.

The Psychological Assessment Battery used are: Multiple Sclerosis Quality of Life-54 (MSQOL-54) scale, Beck Depression Inventory-II, Coping Orientation to Problems Experienced (COPE).

Sample size: The sample consist of patients with MS admitted to the C.A.R.E.N. or Casazza facilities of the IRCCS Centro Neurolesi Bonino-Pulejo in Messina. Twenty eligible subjects recruited and treated with traditional rehabilitation approach plus vibrational therapy. The results will be compared to those obtained from a group of 20 patients who have undergone a traditional rehabilitation treatment without the application of vibrations and who will represent the control group.

A descriptive analysis of the two groups will be performed for clinical and socio-demographic variables. The Shapiro-Wilk test will be applied to assess the distribution of variables. Subsequently, continuous variables will be expressed as mean±sd or median and I-III quartile, while categorical variables in frequency and percentages. An intra-group analysis will be carried out to compare both clinical and instrumental scores between T0 and T1 in each group using either T-Student or Wilcoxon for paired data, and a Pearson correlation or Spearman rank correlation to evaluate the relationship between clinical scales and instrumental data. The inter-group analysis will be applied to compare both clinical and instrumental scores between the groups at T0 and T1 using either a parametric test (T-Student for unpaired data) or a non-parametric test (U-Mann Whitney). The analysis will be performed using the open-source software R3.0. A confidence interval of 95% with a 5% alpha error will be considered. Statistical significance will be set at p<0.05.

The principal investigator (PI) will conduct the study in accordance with good clinical practice (GCP) guidelines and current regulations, and in accordance with the current version of the Declaration of Helsinki.

All study participants will sign informed consent in accordance with current regulations. The study investigator will inform the subject that participation in the protocol is voluntary and that refusal will not in any way affect the relationship with the researcher. Before enrollment in the study, each subject will receive a clear explanation of the nature and purpose of the study from the investigator. A clear information sheet outlining all salient aspects will also be provided in hard copy to the subject, who will have the opportunity to ask any questions and raise any concerns regarding the contents. Additionally, the subject will be given ample time to decide whether to participate in the study before signing the informed consent in duplicate. The original signed informed consent will be retained by the investigator.

Before carrying out any examination provided by this protocol, patients will also provide all authorizations required by law (European Regulation 2016/679, Legislative Decree 196/2003 modified by Legislative Decree no. 101 of 10/08/2018) and by the provisions of the Privacy Guarantor. In accordance with good clinical practice rules, each subject will be uniquely identified by a code, which will be the subject identifier for the entire duration of the studY.

The experimenter will wait for approval from the Ethics Committee. The study in question will be conducted according to the attached protocol, in compliance with the expected timelines, the Declaration of Helsinki (1964 and subsequent amendments), in compliance with Good Clinical Practice guidelines, and in accordance with current regulations.

The study does not involve any additional costs for the institution, nor any external sources of funding of any kind. There is no compensation planned for the study's principal investigator or the involved experimenters. The institution and experimenters are covered by adequate insurance coverage for any damages that may arise from the experimentation.

The proposer agrees to prepare a final report at the conclusion of the study and to make the results publicly available.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of Multiple Sclerosis according to the McDonald criteria;
* Evidence of fatigue symptoms;
* Age between 20 and 60;
* Score on the EDSS scale between 1 and 5.5;
* Signed informed consent.

Exclusion Criteria:

* Pregnancy;
* Presence of cardiac pacemaker or other implants;
* Malignant neoplasms;
* Presence of cardiac, pulmonary, or musculoskeletal comorbidities that contraindicate physical exercise;
* Presence of non-healed wounds;
* Severe visual and/or hearing impairment;

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
mobility | 12 months
  changes in motricity index
postural control | 12 months
  changes in Tinetti's scale
postural control | 12 months
  changes in Berg's scale

SECONDARY OUTCOMES:
fatigue | 12 months
  changes in the Fatigue Severity Scale (FSS)
fatigue | 12 months
  changes in the Modified Fatigue Impact Scale (MFIS)
fatigue | 12 months
  changes in the Fatigue Scale for Motor and Cognitive Functions (FSMC)
fatigue | 12 months
  changes in the Borg Scale
fatigue | 12 months
  changes in the Medical Research Council Scale (MRC)
quality of life | 12 months
  changes in the Multiple Sclerosis Quality of Life-54 (MSQOL-54) scale
quality of life | 12 months
  changes in the Coping Orientation to Problems Experienced (COPE) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Neurolesi Centro Bonino Pulejo, Messina, Sicily, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Formica C, Latella D, Bonanno L, Lombardo Facciale A, Paladina G, Leo A, Pergolizzi L, Fonti B, Quartarone A, Cellini R, Calabro RS. The Role of VibraPlus on Fatigue in Multiple Sclerosis Patients: A Randomized Controlled Trial. J Clin Med. 2025 Jun 5;14(11):3990. doi: 10.3390/jcm14113990. PMID 40507752